CLINICAL TRIAL: NCT00712816
Title: Investigating the Use of a Cryopneumatic Therapy Device in Primary Total Knee Arthroplasty Patients
Brief Title: Use of Cold and Compression Therapy With Total Knee Replacement Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CoolSystems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2007-02
Record Dates: First submitted 2008-07-07; First posted 2008-07-10 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Osteoarthritis; Total Knee Arthroplasty
Keywords: osteoarthritis; total knee arthroplasty; cryotherapy
MeSH Terms: conditions — Osteoarthritis | interventions — Ice

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Device: Game Ready Injury Treatment System (CoolSystems Inc.)
- B (Active Comparator)
  Interventions: Other: Ice with compressive bandages

INTERVENTIONS:
Device: Game Ready Injury Treatment System (CoolSystems Inc.) — Cold with intermittent compression postoperatively for 2 weeks
  Arms: A
Other: Ice with compressive bandages — Cold with static compression postoperatively for 2 weeks
  Arms: B

SUMMARY:
The purpose of the study is to evaluate the effectiveness of a device that delivers cold and intermittent compression as compared to ice and compressive wraps on patients who have undergone knee replacement.

DETAILED DESCRIPTION:
The use of cryotherapy with compression for orthopedic postoperative recovery has not been fully investigated. A new device has been developed that combines cold and intermittent pneumatic compression in a single system. A well-controlled clinical study evaluating the clinical effectiveness of cryotherapy with compression in an orthopedic postoperative application is the subject of this protocol. Patients diagnosed with osteoarthritis of the knee and scheduled for primary total knee arthroplasty procedure will be invited to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 but no more than 85 years of age
* Body Mass Index not greater than 40
* Diagnosis of osteoarthritis of the knee
* Medically cleared for total knee replacement surgery
* Physically and mentally able and willing to participate in and follow the study protocol and schedule
* Able and willing to have all postoperative physical therapy visits in a physical therapy clinic associated with the research site
* Signed informed consent document for the study

Exclusion Criteria:

* Rheumatoid arthritis
* Severe pitting edema in the ipsilateral limb
* History of thrombophlebitis in lower extremities
* An active systemic disease such as AIDS, HIV, hepatitis, etc.
* Is immunologically suppressed or has received or is receiving steroids at any dose daily for more than one month within the last 12 months
* Is pregnant or planning to become pregnant during the study period
* Any condition that would contraindicate using the Game Ready
* Currently enrolled in another clinical trial that could affect outcome of this study
* Previously enrolled in this study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2008-07; Primary Completion 2011-12 (Actual); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Physical function performance | 2 weeks postoperative, 6 weeks postoperative, 6 months postoperative
Time to reach defined physical therapy milestones | 2 weeks postoperative, 6 weeks postoperative, 6 months postoperative

CONTACTS AND LOCATIONS:
Locations (11):
- United States (10):
  - Naval Medical Center, San Diego, San Diego, California
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Central DuPage Hospital, Winfield, Illinois
  - Orthopaedic Research Foundation, Indianapolis, Indiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Hospital for Special Surgery, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Sports Medicine Associates of San Antonio, San Antonio, Texas
  - Madigan Army Medical Center, Tacoma, Washington
- Orthosports, Concord, New South Wales, Australia